CLINICAL TRIAL: NCT07075835
Title: Enhanced External Counterpulsation as a Non-pharmacological Treatment for Patients With Severe and Moderate Ventilation Disorders
Brief Title: Enhanced External Counterpulsation for Patients With Ventilation Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 154247
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Chronic Lung Diseases
Keywords: enhanced external counterpulsation; ventilation disorders; chronic lung diseases; microcirculation; neoangiogenesis; physical activity tolerance
MeSH Terms: conditions — Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main group (Experimental): patients with severe (30% < forced expiratory volume in 1 second < 49% or lung diffusion capacity < 40%) and moderate (50% < forced expiratory volume in 1 second < 59% or lung diffusion capacity 40-60%) ventilation disorders, who are on optimal basic therapy (according to current clinical guidelines) and are in a stable state of respiratory disease (1 month without exacerbation)
  Interventions: Procedure: Enhanced external counterpulsation
- Control group (No Intervention): patients with severe (30% < forced expiratory volume in 1 second < 49% or lung diffusion capacity < 40%) and moderate (50% < forced expiratory volume in 1 second < 59% or lung diffusion capacity 40-60%) ventilation disorders, who are on optimal basic therapy (according to current clinical guidelines) and are in a stable state of respiratory disease (1 month without exacerbation) They will receive only optimal drug therapy for respiratory diseases in accordance with the current clinical guidelines of the Russian Ministry of Health (extended-release beta2-agonists, extended-release m-cholinolytics, inhaled and systemic glucocorticosteroids as needed).

INTERVENTIONS:
Procedure: Enhanced external counterpulsation — 20 (5 days a week for 4 weeks) one-hour procedures (compression pressure 220-280 mmHg) of enhanced external counterpulsation (device: LUMENAIR EECP, Vasomedical Inc., USA, registration certificate №2018/6915 dated 15.03.2018). The systolic deflation/diastolic inflation sequence of enhanced external counterpulsation leads to systolic unloading and diastolic augmentation, resulting in increased blood flow in a pulsatile manner in coronary artery and in others organ arteries.
  Arms: Main group

SUMMARY:
This study evaluates enhanced external counterpulsation as a non-pharmacological therapy for patients with severe and moderate ventilation disorders due to chronic lung diseases (chronic obstructive pulmonary disease, bronchial asthma and interstitial lung diseases). The study will include 80 patients with severe (30% < forced expiratory volume in 1 second < 49% or lung diffusion capacity < 40%) and moderate (50% < forced expiratory volume in 1 second < 59% or lung diffusion capacity 40-60%) ventilation disorders, who will be divided into 2 groups (the main group and the comparison group). In addition to optimal pharmacological therapy according to the current clinical guidelines of the Russian Ministry of Health, the main group will receive a course of enhanced external counterpulsation. The comparison group will receive only optimal pharmacological therapy (according to the current clinical guidelines of the Russian Ministry of Health). At the time of inclusion in the study and after 1 month, spirometry, bodyplethysmography, lung diffusion capacity, a 6-minute walk test and an assessment of quality of life according to the SF-36 questionnaire will be conducted.

DETAILED DESCRIPTION:
Chronic lung diseases represent a significant medical and social burden, leading to reduced quality of life and high disability rates. Despite advances in pharmacotherapy, a subset of patients remains inadequately responsive to pharmacological treatments. Enhanced external counterpulsation, initially developed for cardiology, shows potential for improving pulmonary and respiratory muscle perfusion. This method based on counterpulsation by special cuffs on the legs in the phase of diastole of the heart. The operation of the enhanced external counterpulsation device is synchronized with the patient's electrocardiogram. In the phase of diastole of the heart, there is a rapid sequential inflation of air into the cuffs in the direction from the calves to the buttocks with subsequent compression of arterial vessels and retrograde direction of blood flow in the opposite direction - to the coronary vessels. The cuffs deflate before the next systole. However, its efficacy in pulmonology patients remains understudied. An open-label controlled trial involving 80 patients (n=40 main group, n=40 control group) age 35-74 years with severe (30% < forced expiratory volume in 1 second < 49% or lung diffusion capacity < 40%) and moderate (50% < forced expiratory volume in 1 second < 59% or lung diffusion capacity 40-60%) ventilation disorders, stable condition on optimal therapy (in accordance with the current clinical guidelines of the Russian Ministry of Health (extended-release beta2-agonists, extended-release m-cholinolytics, inhaled glucocorticosteroids, systemic glucocorticosteroids). The main group will receive 20 (5 days a week for 4 weeks) one-hour procedures (compression pressure 220-280 mmHg) of enhanced external counterpulsation (device: LUMENAIR EECP, Vasomedical Inc., USA, registration certificate №2018/6915 dated 15.03.2018) in addition to optimal pharmacological therapy. The comparison group will receive only optimal pharmacological therapy. At the time of inclusion in the study and after 1 month, spirometry (device MIR Spirolab I, bronchodilator 400 mcg of salbutamol - Salbutamol was registered on October 14, 2011, registration number: 001925), bodyplethysmography (Jager Master Screen Body), lung diffusion capacity (Jager Master Screen Body), a 6-minute walk test and an assessment of quality of life according to the SF-36 questionnaire will be conducted. Statistical data processing will be carried out using the StatTech program.

ELIGIBILITY:
Inclusion Criteria:

* Verified severe (30% < forced expiratory volume in 1 second < 49% or lung diffusion capacity < 40%) and moderate (50% < forced expiratory volume in 1 second < 59% or lung diffusion capacity 40-60%) ventilation disorders in patients with different chronic lung diseases who are on optimal basic therapy (according to current clinical guidelines) and are in a stable state of respiratory disease (1 month without exacerbations)
* Signed informed voluntary consent to participate in the study

Exclusion Criteria:

* A history of thrombophlebitis and/or phlebitis
* Thoracic or abdominal aortic aneurysm
* Severe pathology of the valvular heart (Area of orifice in stenoses: Aortic and tricuspid valves: < 1.0 cm²; Mitral valve: < 1.5 cm². Pulmonary valve: pressure gradient between right ventricle and pulmonary artery > 50 mmHg; In case of insufficiency, regurgitation of grade 3-4 according to echocardiography)
* Pregnancy
* High pulmonary hypertension (grade 2-3; >45 mmHg)
* Catheterization cardiac arrest performed within 2-4 weeks before the study
* Tachyarrhythmias (device Myocard-12)
* Uncontrolled arterial hypertension (>180/110 mmHg when treated with 3 drugs, one of which is a diuretic)
* Hemorrhagic conditions critical arterial ischemia of the lower extremities (Stages 3 and 4 of chronic arterial insufficiency of the lower extremities according to the Pokrovsky-Fontaine classification are patients with pain at rest and with trophic or infectious-inflammatory changes in the tissues of the extremities
* Dilatation of the heart cavities (device Philips iU22 Ultrasound)
* Ejection fraction <50% (device Philips iU22 Ultrasound)
* Level of NT-pro BNP > 125 pg/ml
* A history of myocardial infarction
* Severe renal (glomerular filtration rate <30 ml/min/1,73 m2) failure
* Hepatic failure (B and C on the Child-Pugh scale)
* Poor tolerance of the procedure (side effects that disrupt the patient's condition and prevent the continuation of procedures (local: hyperemia, pain, and itching in the area of the cuff application; systemic: hypertensive reaction, dizziness)
* Low patient compliance (skipping more than 3 procedures), refusal to participate in the study
* Exacerbation of the underlying disease during the study

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic of lung volumes | 1 month
  For endpoint the investigators will use bodyplethysmography at the time of inclusion in the study and after 1 month
Dynamic of lung diffusion capacity | 1 month
  For endpoint the investigators will use lung diffusion capacity at the time of inclusion in the study and after 1 month
Dynamic of physical activity tolerance | 1 month
  For endpoint the investigators will use 6-minute walk test at the time of inclusion in the study and after 1 month
Dynamic of quality of life | 1 month
  For endpoint the investigators will use "SF-36 Health Status Survey" questionnaire at the time of inclusion in the study and after 1 month.
  The higher the score, the better the quality of life.

SECONDARY OUTCOMES:
Mortality from all causes | 3 months
  The number of deaths from any cause
Number of hospitalizations due to exacerbation of the underlying disease | 1 months
  Number of hospitalizations for the main disease (chronic obstructive pulmonary disease, bronchial asthma, and interstitial lung diseases)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonology, Clinical Hospital No. 1, I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University)., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
The investigators can't share the research materials because the local ethics committee doesn't allow it.

REFERENCES:
- [Background] Nikolaeva N.A., Lishuta A.S., Voronkova O.O. et al. The Method of Enhanced External Counterpulsation in Clinical Practice. The Russian Archives of Internal Medicine. 2024; 14(5): 339-351. DOI: 10.20514/2226-6704-2024-14-5-339-351. https://www.medarhive.ru/jour/article/view/1850
- [Result] Nikolaeva, N. A. Increase in physical activity tolerance in the background of the use of enhanced external counterpulsation in adult patients with severe respiratory pathology / N. A. Nikolaeva // Modern medicine: the view of a young doctor: Materials of the I International scientific and practical conference for residents and young scientists. In 2 volumes, Kursk, May 16-17, 2023. Volume I. - Kursk: Kursk State Medical University, 2023. - P. 138-140.
- [Result] Nikolaeva N.A., Belenkov Yu.N., Lishuta A.S., Voronkova O.O., Rogova E.F., Buyanova O.E., Abdullaeva G.B. Enhanced external counterpulsation as a measure of non-drug treatment of patients with severe and moderate ventilation disorders. Therapy. 2023; 9(6): 8-14. Doi: https://dx.doi.org/10.18565/therapy.2023.6.8-14